CLINICAL TRIAL: NCT05702957
Title: Letrozole vs Clomiphene Citrate for Induction of Ovulation in Women With Polycystic Ovarian Syndrome: Randomised Control Trial
Brief Title: Letrozole vs Clomiphene Citrate for Induction of Ovulation in Women With Polycystic Ovarian Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Tayyiba Wasim, Professor Obstetrics & Gynaecology, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB/2015/209/SIMS
Record Dates: First submitted 2022-12-08; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: polycystic ovary syndrome; Infertility; Clomiphene citrate; Letrozole
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Letrozole; Clomiphene

STUDY DESIGN:
Intervention Model Description: Total 230 patients were randomized in study, divided in two groups by computer generated numbers, out of which 220 patients were analyzed. .Group-A patients were given clomiphene citrate 50-150mg per day for 5 days starting from 2nd day of menses and group B patients were given letrozole 2.5-7.5mg per day for 5 days.
Who Masked: Participant, Investigator
Masking Description: Two treatment groups were made by random computer generated number i.e. Group A and Group B. Two Concealed boxes labelling A and B containing study drugs were made by pharmacist.Then participants were given drug from concealed boxes according to computer generated number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- letrozole (Experimental): Patients were given letrozole 2.5 mg-7.5mg per day for 5 days started from 2nd day of menses.
  Interventions: Drug: letrozole 2.5mg-7.5mg
- Clomiphene citrate (Active Comparator): Patients were given clomiphene citrate 50-150mg per day for 5 days started from 2nd day of the menses.
  Interventions: Drug: Clomiphene Citrate 50mg-150mg

INTERVENTIONS:
Drug: letrozole 2.5mg-7.5mg — Tab letrozole 2.5 mg-7.5mg per day for 5 days started from 2nd day of menses.
  Other Names: tab lezra 2.5-7.5mg
  Arms: letrozole
Drug: Clomiphene Citrate 50mg-150mg — Tab clomiphene citrate 50-150mg per day for 5 days started from 2nd day of menses.
  Other Names: tab clomid 50-150mg
  Arms: Clomiphene citrate

SUMMARY:
It was randomised controlled study to compare the efficacy of clomiphene and letrozole in polycystic ovarian syndrome(PCOS) women with infertility.The aim was to select more appropriate treatment for ovulation induction in PCOS women.

DETAILED DESCRIPTION:
The prevalence of infertility due to polycystic ovarian syndrome in Pakistan is 21.9%.It leads to an ovulation which results in infertility.The objective of this study was to compare the efficacy of letrozole vs clomiphene citrate for ovulation induction in PCOS women.Methods.It was a randomised controlled trial conducted in department of gynaecology and obstetrics ,Services Hospital Lahore from 2016-2019.

Total 230 patients were included in study, they were divided in two groups, out of which 220 patients were analysed. .Group-A patients were given clomiphene citrate 50-150mg per day for 5 days starting from 2nd day of menses and group B patients were given letrozole 2.5-7.5mg per day for 5 days. Transvaginal ultrasound monitoring done from day 10-12 of menstrual cycle to measure follicle number and size.When follicle achieved a diameter of 18-20mm, then Inj HCG(human chorionic gonadotropin)10,000 IU intramuscular was given. Ovulation was confirmed by day 21 S.progesterone. When patient conceived, they were followed up till delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women age between 18-40 years.
* Normal husband semen analysis.

Exclusion Criteria:

* All infertile couples who had other causes of infertility than PCOS.
* Those who had recently taken these medications.
* Any contraindication to use of drugs e.g renal or hepatic dysfunction, hypersensitivity to this drug.
* BMI>35 because obese women respond poorly to ovulation induction.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 5th week of cycle when periods missed
  Total number of patients conceived after treatment

SECONDARY OUTCOMES:
ovulation rate | 10-22 day of cycle
  when follicle achieved diameter of 18-20mm,HCG given,ovulation confirmed by day 21 progesterone.
Live birth rate | 9 months
  total number of live births divided by total number of patients in a group
Monofollicular development | 10-12 day of menstrual cycle
  when only one follicle achieve diameter of greater than or equal to 18mm
Multifollicular development | 10-12 day of menstrual cycle
  when 2 or more follicles achieve diameter of >12mm
Miscarraige | Less than 24weeks
  spontaneous loss of pregnancy before 24 weeks of gestation
Adverse effects | first 10days of cycle
  hot flushes.
Adverse effects | first 10days of cycle
  Fatigue and dizziness

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical sciences, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Derived] Wasim T, Nasrin T, Zunair J, Irshad S. Efficacy of Letrozole vs Clomiphene Citrate for induction of ovulation in women with polycystic ovarian syndrome. Pak J Med Sci. 2024 Jan-Feb;40(1Part-I):78-83. doi: 10.12669/pjms.40.1.7971. PMID 38196458